CLINICAL TRIAL: NCT02431234
Title: Study of the Mechanisms of the Arterial Calcification of the Members Subordinates in the Diabetes (Implication of the System RANK / RANKL / OSTEOPROTEGERINE)
Brief Title: Arterial Calcification in the Diabetes
Acronym: DIACART
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P111105
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Vascular Diseases; Arteriosclerosis Obliterans; Monckeberg Medial Calcific Sclerosis
Keywords: Type 2 diabetes; Arterial calcification; Mediacalcosis; Calcium score
MeSH Terms: conditions — Diabetic Angiopathies; Arteriosclerosis Obliterans; Monckeberg Medial Calcific Sclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: serum RANKL

SUMMARY:
The blood concentration of the protein RANKL could be predictive of the calcification of the leg arteries, which is a major complication occurring during diabetes. The objective of the DIACART study is to show that blood RANKL concentration predict the progression of calcification of the leg arteries in diabetic patients, independently of other cardiovascular risk factors.

DETAILED DESCRIPTION:
Introduction: Peripheral arterial disease (PAD) is the primary major amputation risk factor in diabetes. The PAD is particularly common among diabetic patients at high cardiovascular risk (20-30% of coronary patients have PAD). The calcification of atherosclerotic plaque and media leg arteries contributes to narrowing of the arterial lumen and exposes the diabetic patient to critical limb ischemia. The receptor RANK (Receptor Activator for Nuclear Factor κ B) and its ligand RANKL form a complex which initially was described as being involved in bone metabolism by activating osteoclasts but the RANK / RANKLigand system could also be involved in the process calcification and arterial obstruction, especially in the lower limbs. Currently there is anti-RANKL antibody used in humans that could possibly slow down this process. But it is necessary to prove the involvement of this system in PAD in diabetic patients at high cardiovascular risk before proposing a therapeutic trial.

Assumptions: the concentration of RANKL could be predictive of calcification of leg arteries in diabetes Main objective: To show that serum RANKL concentrations predict the progression of calcification of the leg arteries in diabetic patients, independently of other cardiovascular risk factors.

Secondary Objectives:

* To show the link between other proteins of bone remodeling, markers of inflammation and glycation, and calcification of leg arteries.
* Measuring the rate of calcification leg arteries.
* Phenotype diabetic patients who have the highest rate of calcification. Primary Outcome: Predictive power of serum RANKL concentration at T0 on the progression of calcification of leg arteries between T0 and T24 months.

Methodology: prospective observational study. The calcium score of leg arteries will be evaluated by a scanner at T0 and 24 months.

Inclusion criteria:

* type 2 diabetes
* women over 60
* men over 50 years
* men and women with known coronary artery disease Non-inclusion criteria:
* severe renal failure
* immunodeficiency
* acute infectious or inflammatory disease
* history of bypass surgery or sub-popliteal angioplasty Number of subjects required: 188 patients will be included. Total study duration: 24 months Inclusion period: 24 months

ELIGIBILITY:
Inclusion criteria:

* type 2 diabetes
* women over 60
* men over 50 years
* men and women with known coronary artery disease

Non-Exclusion criteria:

* severe renal failure
* immunodeficiency
* acute infectious or inflammatory disease
* history of bypass surgery or sub-popliteal angioplasty

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with type 2 diabetes and known coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Serum RANKL concentrations | Baseline
  Serum RANKL concentrations to predict the progression of calcification of the leg arteries in diabetic patients, (independently of other cardiovascular risk factors)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bourron, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetrière, Paris, France

REFERENCES:
- [Derived] Denimal D, Ponnaiah M, Phan F, Jeannin AC, Redheuil A, Salem JE, Boussouar S, Paulstephenraj P, Laroche S, Amouyal C, Hartemann A, Foufelle F, Bourron O. Metabolic dysfunction-associated steatotic liver disease (MASLD) biomarkers and progression of lower limb arterial calcification in patients with type 2 diabetes: a prospective cohort study. Cardiovasc Diabetol. 2025 Apr 23;24(1):176. doi: 10.1186/s12933-025-02705-9. PMID 40269920
- [Derived] Le Goff W, Bourron O, Materne C, Galier S, Phan F, Tan-Chen S, Guillas I, Hartemann A, Salem JE, Redheuil A, Foufelle F, Le Stunff H, Hajduch E, Guerin M. Inverse relationship between circulating sphingosine-1-phosphate and precursor species and coronary artery calcification score in type 2 diabetes. Cardiovasc Diabetol. 2025 Feb 21;24(1):85. doi: 10.1186/s12933-025-02624-9. PMID 39984928
- [Derived] Denimal D, Ponnaiah M, Jeannin AC, Phan F, Hartemann A, Boussouar S, Charpentier E, Redheuil A, Foufelle F, Bourron O. Non-alcoholic fatty liver disease biomarkers estimate cardiovascular risk based on coronary artery calcium score in type 2 diabetes: a cross-sectional study with two independent cohorts. Cardiovasc Diabetol. 2024 Feb 13;23(1):69. doi: 10.1186/s12933-024-02161-x. PMID 38351039
- [Derived] Carlier A, Phan F, Szpigel A, Hajduch E, Salem JE, Gautheron J, Le Goff W, Guerin M, Lachkar F, Ratziu V, Hartemann A, Ferre P, Foufelle F, Bourron O. Dihydroceramides in Triglyceride-Enriched VLDL Are Associated with Nonalcoholic Fatty Liver Disease Severity in Type 2 Diabetes. Cell Rep Med. 2020 Dec 22;1(9):100154. doi: 10.1016/j.xcrm.2020.100154. eCollection 2020 Dec 22. PMID 33377125
- [Derived] Bourron O, Phan F, Diallo MH, Hajage D, Aubert CE, Carlier A, Salem JE, Funck-Brentano C, Kemel S, Cluzel P, Redheuil A, Davaine JM, Massy Z, Mentaverri R, Bonnefont-Rousselot D, Gillery P, Jaisson S, Vermeer C, Lacorte JM, Bouziri N, Laroche S, Amouyal C, Hartemann A. Circulating Receptor Activator of Nuclear Factor kB Ligand and triglycerides are associated with progression of lower limb arterial calcification in type 2 diabetes: a prospective, observational cohort study. Cardiovasc Diabetol. 2020 Sep 18;19(1):140. doi: 10.1186/s12933-020-01122-4. PMID 32948184
- [Derived] Aubert CE, Liabeuf S, Amouyal C, Kemel S, Lajat-Kiss F, Lacorte JM, Halbron M, Carlier A, Salem JE, Funck-Brentano C, Perisic Matic L, Witasp A, Stenvinkel P, Phan F, Massy ZA, Hartemann A, Bourron O. Serum concentration and vascular expression of adiponectin are differentially associated with the diabetic calcifying peripheral arteriopathy. Diabetol Metab Syndr. 2019 Apr 29;11:32. doi: 10.1186/s13098-019-0429-7. eCollection 2019. PMID 31168327